CLINICAL TRIAL: NCT05610254
Title: Rapid Infusion of Ringer's Lactate Solution At Different Temperatures and the Effects on Circulation and Perfusion in Healthy Volunteers - a Randomized Crossover Trial
Brief Title: The Cold Fluids Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); University of Southern Denmark (Other); Simon Fougner Hartmanns Family Foundation (Unknown); Department of Clinical Biochemistry, Vejle Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2022-002137-34
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Hemodynamic Instability
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cold-Warm (Active Comparator): Trial day 1: Participants receive Ringer's lactate cold (15°C, 59°F), Trial day 2: Participants receive Ringer's lactate at body temperature (37°C, 98.6°F)
  Interventions: Drug: Ringer's Lactate
- Warm-Cold (Active Comparator): Trial day 1: Participants receive Ringer's lactate at body temperature (37°C, 98.6°F) Trial day 2: Participants receive Ringer's lactate cold (15°C, 59°F),
  Interventions: Drug: Ringer's Lactate

INTERVENTIONS:
Drug: Ringer's Lactate — On the first trial day healthy volunteers are randomized to receive 30 ml/kg of Ringer's lactate either cold (15°C, 59°F), or at body temperature (37°C, 98.6°F) during a 30-minute interval. After a minimum "washout period" of 24 hours, subjects are switched to receive infusion at the other aforementioned temperatures.

SUMMARY:
In this single center crossover study the aim is to investigate the effect of Ringer's lactate solution at high and low temperatures on physiological response in healthy adults.18 healthy volunteers will be included. Inclusion criteria is; Age between 18-64. Exclusion criteria is; Pre-existing medical problems, Pregnancy (validated through a certified pregnancy test), Body mass index >35 kg/m2, Medication use apart from allergy medication, contraceptives, or non-steroidal anti-inflammatory drugs.

Participants will be randomized to receive 30 ml/kg of Ringer's lactate either cold (15°C, 59°F), or at body temperature (37°C, 98.6°F) during a 30-minute interval. Fluids will be administered through a peripheral vein. After a minimum "washout period" of 24 hours, subjects are switched to receive infusion at the other aforementioned temperatures.

Primary outcome is

* The increase in MAP at 15 minutes after infusion of the fluid bolus. Secondary outcome is
* Time until return of MAP to baseline value after infusion.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-64

Exclusion Criteria:

* Pre-existing medical problems
* Pregnancy (validated through a certified pregnancy test)
* Body mass index >35 kg/m2
* Medication use apart from allergy medication, contraceptives, or non-steroidal anti-inflammatory drugs.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2022-12-03 (Actual); Study Completion 2022-12-03 (Actual)

PRIMARY OUTCOMES:
Increase in MAP at 15 minutes after infusion of the fluid bolus. | 15 minutes

SECONDARY OUTCOMES:
Time until return of MAP to baseline value after infusion. | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biesenbach P, Molmer MB, Svendsen EL, Teichmann D, Wuthe S, Momeni M, Kristensen MR, Laugesen LE, Berg-Beckhoff G, Bentsen LP, Bergmann ML, Brabrand M. Ringer's lactate administered at 15 degrees C leads to a greater and more prolonged increase in blood pressure compared to 37 degrees C. Sci Rep. 2024 Oct 26;14(1):25592. doi: 10.1038/s41598-024-76858-0. PMID 39462030